CLINICAL TRIAL: NCT01038674
Title: A Randomised, Double Blind, Placebo-controlled, Multiple Dose, Dose-escalation, Phase 1 Trial of Anti-IL-20 in Subjects With Rheumatoid Arthritis
Brief Title: Safety and Tolerability of Anti-IL-20 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8226-3704; 2009-013132-20 (EudraCT Number); U1111-1112-6382 (Other: WHO)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-IL-20 (Experimental)
  Interventions: Drug: anti-IL-20
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: anti-IL-20 — Anti-IL-20 injected subcutaneously (under the skin) with 1 dose once weekly during a 6 week period (in total 7 doses) at 2 dose levels.
  Arms: Anti-IL-20
Drug: placebo — Placebo injected subcutaneously (under the skin) with 1 dose once weekly during a 6 week period (in total 7 doses) at 2 dose levels.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety and tolerability of the drug Anti-IL-20 in subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* A diagnosis of rheumatoid arthritis made at least 3 months prior to screening
* Active rheumatoid arthritis, characterised by a DAS28 equal or above 3.2
* Methotrexate treatment (stable dose, equal or below 25 mg/week) for at least 4 weeks prior to study start (subjects receiving stable doses of oral corticosteroids, and/or non-steroidal anti-inflammatory drugs and/or acetaminophen and/or opioids according to prescribed recommended doses can be included)
* Male subjects and female subjects of non-child bearing potential

Exclusion Criteria:

* Body mass index (BMI) less than 18.5 or above 35.0 kg/m2
* Subjects with chronic inflammatory autoimmune disease other than rheumatoid arthritis
* History of or current inflammatory joint disease other than rheumatoid arthritis
* Chronic or ongoing infectious disease requiring systemic anti-infectious treatment within 2 weeks prior to study start
* Past or current malignancy (as judged by the investigator)
* Clinically significant cardiac or cardiovascular disease
* Positive for human immunodeficiency virus (HIV), hepatitis or tuberculosis
* Blood donation or blood loss of more than 0.45L within 2 months prior to study start, or longer if required by local regulations
* Breast-feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | 0 - 21 weeks after dosing

SECONDARY OUTCOMES:
Terminal serum half-life | 0 - 21 weeks after dosing
Maximum observed serum concentration (Cmax) | 6 - 10 weeks after dosing
Change in ACR20, ACR50 and ACR70 | 0-21 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Brussels, Belgium
- Novo Nordisk Investigational Site, Warsaw, Poland

REFERENCES:
- [Result] Lundblad MS, Overgaard RV, Gothberg M, Fjording MS, Watson E. Clinical pharmacokinetics of the anti-interleukin-20 monoclonal antibody NNC0109-0012 in healthy volunteers and patients with psoriasis or rheumatoid arthritis. Adv Ther. 2015 Mar;32(3):228-38. doi: 10.1007/s12325-015-0191-7. Epub 2015 Mar 7. PMID 25749867
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com